CLINICAL TRIAL: NCT06853288
Title: Effects of Ultra Processed Food on Intestinal Energy Harvest
Acronym: UPFEH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: UNC Gillings School of Global Public Health (Unknown)
Responsible Party: Principal Investigator, Faris M Zuraikat, PhD, Assistant Professor of Nutritional Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AAAV3549
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Obesity and Overweight
Keywords: Obesity; Ultra processed Food; Energy balance
MeSH Terms: conditions — Obesity; Overweight | interventions — Food, Processed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 80% Ultra processed (Experimental): Participants will be provided with shopping lists and menus for the two arms of the diet intervention.
  Interventions: Behavioral: Diet containing 80% ultra processed foods
- 20% Ultra processed (Experimental): Participants will be provided with shopping lists and menus for the two arms of the diet intervention.
  Interventions: Behavioral: Diet containing 20% ultra processed foods

INTERVENTIONS:
Behavioral: Diet containing 80% ultra processed foods — Very high ultra-processed food diet where 80% of calories are coming from ultra processed food
  Arms: 80% Ultra processed
Behavioral: Diet containing 20% ultra processed foods — Low ultra processed food diet where 20% of the calories are coming from ultra processed food
  Arms: 20% Ultra processed

SUMMARY:
Ultra processed food is everywhere in modern society and may contain multiple ingredients that affect the way participants' bodies store energy. Some studies have shown that eating a diet high in ultra processed foods leads to weight gain, but these foods have not been studied enough to understand why. Recently, the gut microbiome has become a potential way to measure energy balance in the human body; this is done by measuring how many calories are in the stool. The investigators propose to test a very high ultra-processed food diet where 80% of calories are coming from ultra processed food and a low ultra processed food diet where 20% of the calories are coming from ultra processed food. This study will compare stool sample energy content of the two diets.

DETAILED DESCRIPTION:
This study will recruit people with obesity who are otherwise healthy to participate in this study. Each person will go through baseline testing before starting any of the diets. This consists of one blood draw, one metabolic test which requires each person to remain awake in a small, enclosed room that measures oxygen and carbon dioxide consumption, and one body composition test. Participants will also meet with a study dietitian to review their diet, how to track their diet, and how to collect and ship the stool samples. Each person will be assigned to either 80% or 20% level of ultra processed food in the diet to start and will continue this diet for two weeks. After the first diet phase, each participant will enter a washout period where they will return to eating however they wish and will not need to participate in any research activities. After the two weeks, each participant will return to begin another series of tests and begin the second two-week diet phase. The whole study will take approximately 9 weeks to complete.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-40kg/m2
* weight stable
* able to download app and willing to use it for duration of study
* does own grocery shopping
* otherwise healthy

Exclusion Criteria:

* pregnancy
* history of or planned bariatric surgery
* history of anti obesity medications

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fecal energy loss | 2 weeks
  Amount of calories absorbed from diet will be the difference from energy intake - calories in stool

SECONDARY OUTCOMES:
Microbial taxa | 2 weeks
  Change in types of microbial taxa from baseline to end of diet period

OTHER OUTCOMES:
Insulin, glucose, serum lipid and lipoproteins (mg/dl) | 2 weeks
  Bloods drawn at each timepoint will be assayed for overlapping metabolic markers
C-peptide (ng/ml) | 2 weeks
  Bloods drawn at each timepoint will be assayed for overlapping metabolic markers

CONTACTS AND LOCATIONS:
Overall Officials: Faris M Zuraikat, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Stool samples
Supporting Information: Study Protocol
Time Frame: March 8, 2025 - March 8, 2026

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT06853288/Prot_SAP_001.pdf